CLINICAL TRIAL: NCT06597747
Title: Evaluating Design Improvements With SONNET 3 in Experienced Cochlear Implant Users
Brief Title: Design Improvements With SONNET 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G240188
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SONNET 3 (EAS) (Experimental): Participants complete a take-home trial using SONNET 3 (EAS) audio processor
  Interventions: Device: Audio processor

INTERVENTIONS:
Device: Audio processor — MED-EL SONNET 3 (EAS) audio processor

SUMMARY:
Measuring user-reported satisfaction with the latest behind-the-ear (BTE) audio processor model.

DETAILED DESCRIPTION:
This prospective study will use a single-arm, repeated measures design with subjects serving as their own control. Participants will be experienced cochlear implant (CI) users wearing an approved BTE MED-EL audio processor. Participants will complete a take-home trial with the latest audio processor and then complete a custom questionnaire comparing design and usability to their existing audio processor.

ELIGIBILITY:
Inclusion Criteria:

* Implanted with a MED-EL cochlear implant in at least one ear
* ≥ 12 months since activation of the MED-EL audio processor
* Consistently using a SONNET (EAS) or SONNET 2 (EAS) Audio Processor
* Ability to complete all study procedures
* Participant and parental (if applicable) commitment to comply with all study procedures for the duration of the study

Exclusion Criteria:

* Evidence that hearing loss is retrocochlear in origin
* Unable to provide reliable feedback during cochlear implant programming
* Skin or scalp condition precluding use of the study device
* Unrealistic participant or parent (if applicable) motivation or expectations
* Participants without a stable fitting map at enrollment e.g., due to changes in hearing, global health status, etc.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-16 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Group level results will be reported.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SONNET 3 (EAS)
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SONNET 3 (EAS)
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (24.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  United States | 20
Cochlear Implant Experience [Mean (Standard Deviation); unit: years] — Years since activation of cochlear implant
  years | 6.1 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Participants Reporting Improvement With SONNET 3 Design
Description: The proportion of participants reporting improvement in design aspects of SONNET 3 (EAS) on a user survey
Time Frame: Measured 1 month after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | SONNET 3 (EAS)
Number analyzed (Participants) | 20
Participants | 20

2. Secondary Outcome: Audiologist Satisfaction Ratings
Description: Score on a 6-point Likert scale (1 = Strongly Disagree to 6 = Strongly Agree; higher scores indicate better outcomes). Values reported are the average scores on subsections of the audiologist survey.
Time Frame: Measured after study completion, an average of 7.5 months
Measure: Mean (Standard Deviation); unit: Score on 6-point Likert scale
Groups:
- Audiologist: Audiologists who programmed the SONNET 3 (EAS) for the study completed a survey on their experience at the conclusion of the study.
Arm/Group | Audiologist
Number analyzed (Participants) | 3
Score on 6-point Likert scale
  SONNET 3 Design | 5.4 (0.3)
  MAESTRO 11 | 5.5 (0.5)

ADVERSE EVENTS:
Time Frame: Measured through study completion, an average of 7.5 months
Arm/Group | SONNET 3 (EAS)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SONNET 3 (EAS) (N=20)
Adverse Device Effect (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-02): https://cdn.clinicaltrials.gov/large-docs/47/NCT06597747/Prot_SAP_000.pdf